CLINICAL TRIAL: NCT04978064
Title: E-health Psychological Intervention in Pregnant Women Exposed to Intimate Partner Violence (eIPV): a Pilot Randomised Controlled Trial
Brief Title: E-health Psychological Intervention in Pregnant Women Exposed to Intimate Partner Violence (eIPV)
Acronym: eIPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: University of Southern Denmark (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Antonella Ludmila Zapata Calvente, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: eIPV; 202167133116 (Other: Andalusian Research Ethics Committee); 20212000-80 (Other: Regional Committees Health Research Ethics Southern Denmark)
Record Dates: First submitted 2021-07-04; First posted 2021-07-27 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Pregnancy Related; Violence, Gender-Based; Intimate Partner Violence
Keywords: pilot randomized controlled trial; pregnancy; intimate partner violence; e-health intervention; counselling

STUDY DESIGN:
Intervention Model Description: A pilot randomised controlled trial (RCT), co-designed by patient input using a modified Zelen's design with additional qualitative evaluation, will be nested within a cohort study.
Who Masked: Participant
Masking Description: Women in the intervention group will be blinded but not women in the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Behavioral e-health psychological counselling
  Interventions: Behavioral: e-health psychological counselling
- Control group (Other): Usual care (delayed behavioral e-health psychological counselling)
  Interventions: Behavioral: e-health psychological counselling

INTERVENTIONS:
Behavioral: e-health psychological counselling — Intervention group: Women positive for IPV who accept the e-Health intervention and who have been randomly allocated in the intervention group will receive the e-health package as the rest of the cohort, as well as the baseline and outcome measurements. The e-health package will include six video counselling sessions by trained providers and the access to a mobile application for designing security plans, an adapted version of the mobile application "My Plan". The content of the six individually tailored sessions will be based on the Dutton's Empowerment Model and the Psychosocial Readiness Model.
  Control group: women positive in IPV who accept the e-Health intervention package will be asked for a second consent to receive a delayed intervention (8 weeks later) and to complete as the baseline and outcome measurements. Women can request to leave the control group at any time and to receive the intervention immediately (in which case they data will be part of the cohort study).

SUMMARY:
The investigators will assess the need and feasibility of randomising a sufficiently large number of women exposed to IPV during pregnancy in a full-scale future randomised trial. To achieve this, the investigators will:

1. estimate rates of consent to randomization, and the rates of adherence and dropout following randomization (for the use in sample size estimation)
2. determine recruitment duration
3. examine the women's perception about the benefit of the intervention
4. determine the reasons for acceptability, non-adherence, and obstacles to recruitment, randomisation and consent through qualitative interviews

DETAILED DESCRIPTION:
Introduction. Intimate partner violence (IPV) during pregnancy, a condition as common as obstetrics conditions like gestational diabetes, is associated with maternal and neonatal complications. Systematic detection of IPV is not well established in antenatal screening probably because the effectiveness of protective interventions has not been evaluated. Among mothers exposed to IPV, e-health interventions during pregnancy may be beneficial. Prior to performing a full-scale effectiveness trial for such an intervention, a pilot study is required to assess the need and feasibility of randomising a sufficiently large number of women at exposed to IPV during pregnancy.

Methods. The eIPV trial is a randomised pilot study nested within a cohort of consenting mothers at <12 weeks' gestation who screen positive for IPV in the first antenatal visit and accept an e-health package (psychological counselling by videoconference) in Spain and Denmark. Twenty eligible mothers from the above cohort will be randomised to either intervention or control. The intervention group will receive the e-health package as part of the cohort. The control group will be invited to accept a delay in the intervention (e-health package eight weeks later). After consenting to delay, the control group will provide comparative data without losing the opportunity of obtaining the intervention. The investigators will determine estimates of rates of informed consent to randomization, and the rates of adherence and dropout following randomization. Qualitative interviews will be conducted to examine the women's perception about the benefit of the intervention, reasons for acceptability and non-adherence, and obstacles to recruitment, randomisation and consent. The results will inform the feasibility and variance of key clinical outcome measures for estimation of sample size of the full-scale effectiveness trial.

Comment. The pilot study nested within the cohort study will allow us to obtain information about the rates of IPV in pregnancy, the acceptability of an e-health intervention and the availability of participants for randomisation into a large effectiveness trial.

ELIGIBILITY:
Inclusion Criteria:

• Pregnant women at <12 weeks gestation, who screen positive in IPV at the first antenatal visit and accept the e-health package.

Exclusion Criteria:

* Women who cannot be informed about the study without their partners or other family members knowing
* Women mentally or physically incapacity to participate in the study
* Women below 16 years in Spain or below 18 years in Denmark
* Inability to understand Danish/Spanish
* Lack of internet and electronic device
* Women with extreme severity of IPV. Women selected to participate in the trial in this situation will receive a danger assessment before randomisation and if the severity of IPV is confirmed, they will be routinely treated and supported according to the standard protocol in each country. Women who have same-sex partners will be screened, but their data will not be used for the purpose of this study.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Consent rate for a future full-scale RCT trial | Three to nine months
  Rate of women who were positive in IPV, consent to receive e-health package and consent to randomization in the control group.

SECONDARY OUTCOMES:
Positivity rate of the cohort study (useful for planning the future full-scale randomised control trial): | Three to nine months
  Rate of women who were positive in IPV and consent to receive e-health package
Completion rate in the intervention group a future full-scale RCT trial | Three to nine months
  Rate of women who were recruited to intervention group, and for whom complete outcomes were obtained.
Completion rate in the control group a future full-scale RCT trial | Three to nine months
  Rate of women who were recruited to control group, and for whom complete outcomes were obtained.
Recruitment duration for a future full-scale RCT trial | Three to nine months
  Recruitment duration (in days) to get the pilot sample (5 women for the intervention group and 5 women for the control group, in each country)
Benefit of the intervention a future full-scale RCT trial | Three to nine months
  Perception of the intervention by women participating in the pilot through the information obtained in qualitative interviews.
Perception about the delay of the intervention of the control group for a future full-scale RCT trial | Three to nine months
  Perception about the duration of delay of the intervention of women in the control group (provided in the qualitative interviews).
Reasons for acceptability, non-adherence, and obstacles for a future full-scale RCT trial | Three to nine months
  Reasons for acceptability, non-adherence, and obstacles to recruitment, randomization, consent and follow-up (provided in the qualitative interviews).
Follow up rate for a future full-scale RCT trial | Three to nine months
  Rate of failure to obtain data in the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Khalid S. Khan, Study Director — Universidad de Granada
Locations (2):
- Odense University Hospital, Odense, Denmark
- University of Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Yes
We will collaborate in an approved, registered Individual Participant Data metaanalysis
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Starting 6 months after publication
Access Criteria: On reasonable request, protocol, data collection forms and published results are available from investigators. Sharing would need to be comply with data protection laws.

REFERENCES:
- [Background] Martin-de-Las-Heras S, Velasco C, Luna-Del-Castillo JD, Khan KS. Breastfeeding avoidance following psychological intimate partner violence during pregnancy: a cohort study and multivariate analysis. BJOG. 2019 May;126(6):778-783. doi: 10.1111/1471-0528.15592. Epub 2019 Jan 24. PMID 30575266
- [Background] Roman-Galvez RM, Martin-Pelaez S, Martinez-Galiano JM, Khan KS, Bueno-Cavanillas A. Prevalence of Intimate Partner Violence in Pregnancy: An Umbrella Review. Int J Environ Res Public Health. 2021 Jan 15;18(2):707. doi: 10.3390/ijerph18020707. PMID 33467538
- [Background] Rasch V, Van TN, Nguyen HTT, Manongi R, Mushi D, Meyrowitsch DW, Gammeltoft T, Wu CS. Intimate partner violence (IPV): The validity of an IPV screening instrument utilized among pregnant women in Tanzania and Vietnam. PLoS One. 2018 Feb 1;13(2):e0190856. doi: 10.1371/journal.pone.0190856. eCollection 2018. PMID 29389954